CLINICAL TRIAL: NCT05552248
Title: Assessment of the Safety and Performance of a Lumbar Belt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Decathlon SE (Industry)
Collaborators: EFOR, France (Industry)
Responsible Party: Sponsor
Other Study IDs: lumbarSOFT300-MID500
Record Dates: First submitted 2022-09-13; First posted 2022-09-23 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Orthosis group 1: Use of LumbarBelt Soft 300 device during sport practice (for 12 weeks)
  Interventions: Device: LumbarBelt SOFT 300
- Control group 1: Control group of the LumbarBelt Soft 300 group - no medical device used during sport practice (for 12 weeks)
  Interventions: Other: Control group LumbarBelt SOFT 300
- Orthosis group 2: Use of LumbarBelt Mid 500 device during sport practice (for 12 weeks)
  Interventions: Device: LumbarBelt MID 500
- Control group 2: Control group of the LumbarBelt Mid 500 group - no medical device used during sport practice (for 12 weeks)
  Interventions: Other: Control group LumbarBelt MID 500

INTERVENTIONS:
Device: LumbarBelt SOFT 300 — 15 patients will be included in this group and will used the medical device LumbarBelt SOFT 300 during sport practice (at least 2 sport sessions per week), for 12 weeks.
  Groups: Orthosis group 1
Other: Control group LumbarBelt SOFT 300 — 15 patients will be included in this control group and will performed their sport sessions as usual (without the medical device LumbarBelt SOFT 300), for at least 2 sport sessions per week during 12 weeks.
  Groups: Control group 1
Device: LumbarBelt MID 500 — 15 patients will be included in this group and will used the medical device LumbarBelt MID 500 during sport practice (at least 2 sport sessions per week), for 12 weeks.
  Groups: Orthosis group 2
Other: Control group LumbarBelt MID 500 — 15 patients will be included in this control group and will performed their sport sessions as usual (without the medical device LumbarBelt MID 500), for at least 2 sport sessions per week during 12 weeks.
  Groups: Control group 2

SUMMARY:
Decathlon has developed the Lumbar belt Soft 300 and Mid 500 products which are medical devices designed to reduce pain and improve function during sport practice for athletes with a common subacute or chronic low back pain.

The objective of this multicentre study is to collect data on the related clinical complications and clinical outcomes of market-approved Decathlon Lumbar belt range of products to demonstrate safety and performance of these devices in a real-world setting.

Outcome data collected from this study will provide the basis for Post-Market Surveillance (PMS) reporting, Clinical Study Report (CSR), Clinical Evaluation Report (CER) on Decathlon lumbar belt Soft 300/ Mid 500 devices and support peer-reviewed publications on products performance and safety.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥18 years old
* Subject has a medically-confirmed common subacute or chronic low back pain
* Subject performs regular physical activity
* The current condition of his/her back allows the subject to pursue a usual physical activity
* Subject has been informed and is willing to sign an informed consent form
* Subject is willing to comply with protocol requirements and return to the study center for all clinical evaluations and required follow-up (12 weeks)
* Subject is affiliated to the French social security regime

Exclusion Criteria:

* Subject has undergone a surgical treatment for his/her back
* Subject presents associated neurologic signs (equina syndrome, radiculopathy, sciatica…)
* Subject presents signs of specific low back pain (i.e. low back pain is a symptom of an underlying condition): presence of red flags
* Subject has conditions that may interfere with his/her ability to understand protocol requirements, participate in scheduled visits, or provide his/her informed consent
* Subject has worn a support (lumbar or sacroiliac hip belt) during sports sessions in the last month
* Subject has any medical condition that could impact the study at investigator's discretion
* Subject has a known hypersensitivity or allergy to the components of the devices (elastodiene, elastane, polyamide, polyethersulfone [PES])
* Adult subject to a legal protection measure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with medically-confirmed common subacute or chronic low back pain whose current condition of his/her back allows the subject to pursue a usual physical activity.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Functionnal score | Change from Baseline functionnal score at 12 weeks
  Comparison of the Oswestry Disability Index (10-item questionnaire with a global score from 0=best outcome to 100=worst outcome) between the baseline and last follow-up visit in each group (orthosis vs control), for each device model

SECONDARY OUTCOMES:
Confidence level (confidence questionnaire related to physical activity) | Change from Baseline confidence level at 12 weeks
  Gap in the confidence level related to physical activity (scale from 0=worst outcome to 100=best outcome), between the baseline and last follow-up visit in each group (orthosis vs control), for each device model
Low back pain | Change from Baseline low back pain at 12 weeks
  Comparison of low back pain, assessed through a Numerical Rating Scale (NRS) ranging from 0=best outcome to 10=worst outcome, between the groups (orthosis vs control), for each device model
Safety (adverse events) | 12 weeks of follow-up
  Comparison of adverse events rates between the groups (orthosis vs control), for each device model

CONTACTS AND LOCATIONS:
Overall Officials: Yoann MORVAN, Principal Investigator — Boulogne sur Mer Hospital Center
Locations (2):
- France (2):
  - Centre Hospitalier de Boulogne-sur-Mer, Boulogne-sur-Mer
  - Centre de rééducation et de balnéothérapie Kinés Faches, Faches-Thumesnil

IPD SHARING:
Plan to Share IPD: No